CLINICAL TRIAL: NCT04392271
Title: Assessment of Brain O-GlcNAcase (OGA) Enzyme Occupancy After Multiple Oral Doses of LY3372689 as Measured by Positron Emission Tomography (PET) With the Radioligand [18F]LY3316612 in Healthy Subjects
Brief Title: A Study of the Effects of Multiple Doses of LY3372689 on the Brain in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17243; I9X-MC-MTAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-04-21; First posted 2020-05-18 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3372689 + [18F]LSN3316612 (Experimental): LY3372689 administered orally followed by [18F]LSN3316612 PET tracer administered intravenously (IV) approximately 24 hours later.
  Interventions: Drug: LY3372689; Diagnostic Test: [18F]LSN3316612

INTERVENTIONS:
Drug: LY3372689 — Administered orally.
Diagnostic Test: [18F]LSN3316612 — Administered intravenously (IV).
  Other Names: [18F]MNI-1068

SUMMARY:
This study uses imaging to evaluate how LY3372689 binds to a protein in the brain. This study will be conducted in healthy participants and will last up to about 10 weeks. Screening must be completed within four weeks prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females who do not have child-bearing potential
* Have a body mass index (BMI) of greater than (>)18 to less than or equal to (≤32) kilograms per square meter (kg/m²), inclusive, at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG, heart tracing), blood and urine laboratory test results that are acceptable for the study
* Have venous access sufficient to allow for blood sampling

Exclusion Criteria:

* Have a history of head injury or contraindications to undergoing magnetic resonance imaging (MRI) examination
* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have had prior participation in other research protocols or clinical care in the preceding year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure exceeds the effective dose of 50 milliSievert (mSv), which would be above the acceptable annual limit established by the US Federal Guidelines
* Are current smokers or have used tobacco or nicotine-containing products as determined by the cotinine test
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate or could interfere with understanding the results of the study
* Participate in regular vigorous exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Percent O-GlcNAcase (OGA) Enzyme Occupancy (EO) | Approximately 2 to 96 hours following the first dose
  Percent OGA EO
Percent OGA EO | Approximately 2 to 96 hours following the last dose
  Percent OGA EO

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve During the Dosing Interval (AUC[0-tau]) of LY3372689 | Baseline through 24 hours
  PK: AUC(0-tau) of LY3372689
PK: Maximum Concentration (Cmax) of LY3372689 | Baseline through 24 hours
  PK: Cmax of LY3372689

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No